CLINICAL TRIAL: NCT03925168
Title: Music Therapy and Dialysis: A Pilot Investigation Into the Effectiveness of Patient-Selected Music Interventions on Physiological, Psychological, and Quality-of-Life Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tulane University (Other)
Collaborators: National Kidney Foundation, United States (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-866
Record Dates: First submitted 2019-04-16; First posted 2019-04-24 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: End Stage Renal Disease; Depression; Anxiety; Major Depressive Disorder; Generalized Anxiety Disorder; Compliance, Patient; Compliance, Medication; Mood; Pain; Energy Supply; Deficiency; Quality of Life; Blood Pressure; Heart Rate Fast
Keywords: end stage kidney disease; depression; major depressive disorder; anxiety; generalized anxiety disorder; music therapy; dialysis; quality of life; blood pressure; heart rate; pain; energy; mood; medication compliance; music
MeSH Terms: conditions — Kidney Failure, Chronic; Depression; Anxiety Disorders; Depressive Disorder, Major; Generalized Anxiety Disorder; Patient Compliance; Medication Adherence; Pain; Tachycardia | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: Cluster-randomized clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Music therapy
  Interventions: Behavioral: Music therapy
- Control (No Intervention): No music therapy

INTERVENTIONS:
Behavioral: Music therapy — Music therapy will be administered according to the Eyre (2008) decision tree model. According to this model, the patient chooses his or her preferred musical intervention at the beginning of each session. Choices include: sing songs, compose a song, listen to songs, play instruments, have an imagery experience, listen to music, improvise, and use music for relaxation.
  Arms: Experimental

SUMMARY:
The objective of this study is to determine the effect of music therapy during dialysis on:

depression, anxiety, quality of life, blood pressure, heart rate, medication compliance, compliance with dialysis treatment, number of hospitalizations, pain level, and energy level.

DETAILED DESCRIPTION:
This study will be a cluster-randomized clinical trial. In order to limit contamination bias, dialysis sessions at each site will be randomized to the experimental group or the wait-list control group. For example, patients receiving MWF first-session dialysis may be randomized to the experimental group while patients receiving TTS second-session dialysis may be randomized to the control group. Due to this randomization scheme, patients will be able to receive individualized music therapy while sitting in an open dialysis unit. The subject population includes English-speaking, adult (21+) hemodialysis patients who receive dialysis at the one of the two outpatient dialysis centers included in this study. Subjects will be excluded if they do not speak English or if they are deaf as these patient populations would not be likely to benefit from music therapy administered in English. Up to 100 patients will be enrolled in this study.

Patients receiving dialysis at DCI, Inc, who consent to participate and are randomized to the experimental group will receive 30-minute music therapy sessions over the course of several months. Music therapy will be administered by certified music therapists and music therapy students according to the Eyre (2008) decision tree model. According to this model, the patient chooses his or her preferred musical intervention at the beginning of each session. Choices include: sing songs, compose a song, listen to songs, play instruments, have an imagery experience, listen to music, improvise, and use music for relaxation. If the patient is unwilling or unable to make a decision, then the music therapist will choose an intervention based on the patient's perceived needs. For example, if the perceived need is expression of emotions, then the music therapist may suggest song composition, song choice, song singing, or improvisation. The music therapist will continue to assess the client's perceived needs based on their physical, verbal, and emotional responses to the chosen musical interventions, and the therapist will adjust their musical interventions accordingly (the complete Eyre Decision Tree Model is attached). The instruments utilized in music therapy will include a classic guitar, gato box (a small, drum-like instrument), and a 3-piece egg shaker set. All of these instruments can be played loudly enough to provide music therapy to the patient but softly enough as to not disturb the adjacent patients in the dialysis unit. In fact, these instruments are frequently used to provide music therapy to patients in open neonatal intensive care units.

The primary variables in this study include depression, anxiety, and quality of life. The median time to recovery for a major depressive episode is 20 weeks; therefore, patients randomized to the control group will receive music therapy for approximately 20 weeks. Depression will be measured using the Patient Health Questionnaire-9 (PHQ-9), anxiety will be measured using the Generalized Anxiety Disorder-7 (GAD-7), and quality of life will be measured using the Kidney Disease and Quality of Life (KDQOL™-36) questionnaire. These tools are self-administered questionnaires that will be provided by the music therapists to both the experimental and control groups once a month during the study. Any patient with a PHQ-9 score greater than 10 (moderate depression) or a GAD-7 score greater than 10 (moderate anxiety) will additionally be given resources for available mental health providers in the area. While these tools are validated to be utilized every two weeks, they will be utilized every month during this study to limit testing fatigue. In addition, the PHQ-9, GAD-7, and KDQOL™-36 will be administered 30, 60, and 90 days after the experimental group receives their last music therapy session to both the experimental and control groups to assess for recurrent episodes. Among patients with major depressive disorder, recurrent episodes occur in approximately 50 percent. The risk of reoccurrence appears to be greatest in the first few months after cessation of depressive therapy.

The secondary variables in this study include blood pressure, heart rate, medication compliance, compliance with dialysis treatment, number of hospitalizations, pain level, and energy level. The music therapists will record the heart rate (HR) and blood pressure (BP) of each patient at the beginning of dialysis as well as at the beginning and end of music therapy (or a 30-minute period during which music therapy would have been administered). These HRs and BPs will be recorded using nursing vitals. Prior to the start of each session, the music therapist will provide self-administered questionnaires that ask patients to rate their pain (utilizing the Numeric Rating Scale [NRS-11]), mood, anxiety, and energy level. The patients will rate their pain, mood, anxiety, and energy level at the end of the session as well. The music therapist will record if the patient stayed for their entire treatment, or if they asked to stop dialysis early (the complete weekly and monthly data collection forms are attached). Music therapy sessions will be audio recorded using a condenser microphone and iPad Pro, and any subjective feedback from dialysis patients about music therapy sessions will be recorded as well.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking, adult (21+) hemodialysis patients who receive dialysis at the one of the two outpatient dialysis centers

Exclusion Criteria:

* do not speak English, deafness

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-03-08 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Depression | Until 90 days post study
  Measured by Patient Health Questionnaire 9 (PHQ-9). The PHQ-9 measures depression symptoms. Scores range from 0 to 27. A score of 0 to 4 indicates no depression symptoms, 5 to 9 indicates mild symptoms, 10 to 14 indicates moderate symptoms, 15 to 19 indicates moderately severe symptoms, and 20 to 27 indicates severe symptoms.
Anxiety | Until 90 days post study
  Measured by Generalized Anxiety Disorder 7 patient screening tool (GAD-7). The GAD-7 measures anxiety symptoms. Scores range from 0 to 21. A score of 5 or higher indicates mild anxiety, 10 or higher indicates moderate anxiety, and 15 or higher indicates severe anxiety.
Measuring change in Quality of life using Kidney Disease and Quality of Life 36 patient screening tool (KDQOL36) | Until 90 days post study
  Measured by Kidney Disease and Quality of Life 36 patient screening tool. The KDQOL36 measures quality of life for kidney disease patients. Scores range from 36 to 172. Lower scores indicate greater quality of life. Appropriate scores vary by age.
Compliance with dialysis | Up to 5 months
  Self-reported
Number of hospitalizations | Up to 5 months
  Self-reported

SECONDARY OUTCOMES:
Blood pressure | Up to 5 months
Heart rate | Up to 5 months
Medication compliance questionnaire. | Up to 5 months
  A questionnaire about medication compliance will be administered to patients so that they can self report compliance with medications and compliance with dialysis.
Measure change in Pain using the Numeric Rating Scale 11 (NRS11) | Up to 5 months
  Measured by the Numeric Rating Scale 11. This scale ranges from 0 to 11. A score of 0 indicates no pain while a score of 11 indicates severe pain.
Participant Energy | Up to 5 months
  A questionnaire about energy will be administered to patients so that they can rate their energy on a scale from 0 to 5. A score of 0 indicates no energy while a score of 5 indicates a great amount of energy.
Mood | Up to 5 months
  A questionnaire about mood will be administered to patients so that they can rate their mood on a scale from 0 to 5. A score of 0 indicates poor mood while a score of 5 indicates a great mood.

CONTACTS AND LOCATIONS:
Overall Officials: Angelina Dixon, MD, Principal Investigator — Tulane University
Locations (3):
- United States (3):
  - DCI Canal Street, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - DCI West Bank, Terrytown, Louisiana

IPD SHARING:
Plan to Share IPD: No